CLINICAL TRIAL: NCT03770273
Title: A Phase 2 Randomized Double-Blinded Placebo-Controlled Study to Evaluate the Safety and Efficacy of Subcutaneous Sarilumab in Improving the Quality of Life in Subjects With Indolent Systemic Mastocytosis
Brief Title: Safety and Efficacy of Subcutaneous Sarilumab in Improving the Quality of Life in People With Indolent Systemic Mastocytosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 190027; 19-I-0027
Record Dates: First submitted 2018-12-07; First posted 2018-12-10 (Actual); Results first posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2023-08-24

CONDITIONS: Indolent Systemic Mastocytosis
Keywords: Cytokine; Monoclonal Therapy; Interleukin-6; Mast Cell; Bone Marrow
MeSH Terms: conditions — Mastocytosis, Systemic | interventions — sarilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Drug: sarilumab (Active Comparator): Participants with indolent systemic mastocytosis receive sarilumab 200 mg (1.14 ml) subcutaneous injection every two weeks for 16 weeks (8 doses total)
  Interventions: Biological: sarilumab
- Placebo (Active Comparator): Participants with indolent systemic mastocytosis receive placebo subcutaneous injection every two weeks for 16 week (8 doses total)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: sarilumab — Sarilumab is a fully human anti-IL-6Rα monoclonal antibody that binds membrane-bound and soluble human IL-6R and has been shown to inhibit IL-6 signaling.
  Arms: Drug: sarilumab
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Background:

Mast cells help the body fight disease and heal wounds. People with indolent systemic mastocytosis (ISM) make too many mast cells. This causes pain, tiredness, digestive problems, and other symptoms. Researchers think the drug sarilumab could help.

Objective:

To see if sarilumab is a safe and effective treatment for people with ISM.

Eligibility:

Adults ages 18-75 with ISM who are enrolled in NIH study 02-I-0277

Design:

Participants will be screened with:

* Physical exam
* Medical history
* Blood and urine tests
* Questionnaires
* Bone marrow removed by a needle inserted into the hip bone
* Ultrasound of the abdomen
* Photographs of the skin

Participants will repeat some screening tests at study visits.

Participants will have a baseline visit in the hospital for 3 days. They will:

* Be assigned to get either the study drug or a placebo. They will not know which one they get.
* Have a skin punch biopsy: An instrument will remove a small piece of skin.
* Get their first drug dose injected under their skin

Participants will keep a side effect and medication diary during the study.

Participants will visit the clinic to get a drug dose every 2 weeks, for a total of 8 doses.

Participants will have a visit 2 weeks after their final dose. It will last up to 2 days.

Participants will have another visit 12 weeks later.

Participants may then continue this study for 1 more year. Those who continue will get sarilumab, even if they previously got the placebo, every 2 weeks. They will have visits every 6 weeks, and then every 3 months.

DETAILED DESCRIPTION:
Systemic mastocytosis is a disorder caused by clonal mast cell proliferation and release of mast cell mediators including tryptase. As a result, mast cell numbers may increase and affect target organs including the dermis (maculopapular cutaneous mastocytosis/urticaria pigmentosa, flushing), gastrointestinal tract (abdominal pain, diarrhea), skeletal system (osteoporosis), hematological system (anemia, thrombocytopenia), and spleen and liver (organomegaly). Patients with indolent (non-aggressive) systemic mastocytosis (ISM) are not candidates for cytoreductive therapy and are generally treated with symptomatic therapy that only partly decreases symptoms. There is, however, a documented association between severity of mastocytosis and elevated serum levels of interleukin (IL)-6. Furthermore, mast cells have been shown to double their rate of division and exhibit increased reactivity and release of mediators when cultured in the presence of IL-6. In addition, in an animal model of mastocytosis, anti-IL-6 has been shown to slow disease progression. In this study, adults with ISM will thus be randomized and treated with sarilumab, a recombinant monoclonal antibody directed against the IL-6 receptor, or receive placebo. Sarilumab is marketed in the United States as Kevzara (Sanofi/Genzyme [Cambridge, Massachusetts, USA ]) and is approved by the Food and Drug Administration for the treatment of rheumatoid arthritis. Binding of sarilumab to the IL-6 receptor inhibits IL-6-associated human mast cell signaling and proliferation with a resultant decrease in proliferation and reactivity (decreased mediator release), and therefore is a rational choice for the treatment of ISM.

In this study, participants will be randomized with approximately half of the participants receiving study drug, which will be administered at 200 mg via subcutaneous (SC) injection once every 2 weeks (Q2W) for a total of 16 weeks. The other participants will receive a placebo administered via SC injection Q2W for 16 weeks. Participants will return for a follow-up visit 2 weeks after the final dose (treatment peak), and then again 12 weeks later. Evaluations at study visits will include quality of life and symptom assessments and measurement of serum tryptase levels. Bone marrow examination will be performed at the onset and conclusion of the study. After the week 28 visit, all participants will have the option to continue sarilumab for 52 more weeks, at 200 mg administered via SC injections. Participants will continue to be monitored on a regular basis for safety concerns, as instructed in the study drug s package insert.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants must meet all of the following criteria to be enrolled in this study:

1. Male or female participant greater than or equal to 18 and < 75 years of age at screening.
2. Enrolled on NIAID protocol 02-I-0277.
3. Documented pathologic diagnosis of ISM.
4. Mc-QoL score of at least 25% (which suggests participant is at least somewhat affected by all Mc-QoL questions).
5. Willing and able to undergo a bone marrow biopsy and aspirate.
6. Absolute neutrophil count (ANC) greater than or equal to 2000/mL.
7. Hemoglobin greater than or equal to 12.0 g/dL (males), greater than or equal to 11 g/dL (females).
8. Platelet count greater than or equal to 150,000/microliters.
9. Alanine transaminase (ALT) and aspartate transaminase (AST) < 1.5 times the upper limit of normal (ULN).
10. Willing to allow storage of blood and bone marrow for future use in medical research.
11. Willing to allow genetic testing on biospecimens.
12. Able to provide informed consent.
13. Participants who can become pregnant must agree to use adequate contraception when engaging in sexual activities that can result in pregnancy. Adequate contraception must be used consistently, beginning at least 1 month before the beginning of dosing and lasting until 3 months after the final dose of study drug. Acceptable methods of contraception include the following:

    * Hormonal contraception (non-oral only).
    * Male or female condom with spermicide.
    * Diaphragm or cervical cap with a spermicide.
    * Intrauterine device.

EXCLUSION CRITERIA:

Individuals meeting any of the following criteria will be excluded from study participation:

1. Any abnormality that would be scored as a Grade 4 toxicity on the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Only clinically significant lab results will deem the subject ineligible
2. Infected with HIV or has other known immunodeficiency.
3. Has an active infection, including localized infection.
4. Active diverticulitis.
5. Active or chronic viral hepatitis.
6. Active or latent tuberculosis.
7. Use of any other anti-IL-6 or anti-IL-6R agent within 1 year prior to the date informed consent was obtained.
8. Use of cytoreductive therapy for mastocytosis within 1 year prior to the date informed consent was obtained.
9. Known lymphoma or advanced and metastatic solid tumors on active therapy (including chemotherapy) within 1 year prior to the date informed consent was obtained
10. Use of chemotherapy within 1 year prior to the date informed consent was obtained.
11. Receipt of any marketed (eg, omalizumab) or investigational biologic or monoclonal antibody reported to affect mast cell activation within 5 half-lives prior to date informed consent was obtained.
12. Receipt of intravenous (IV) immunoglobulin within 30 days prior to the date informed consent was obtained.
13. Receipt of live attenuated vaccines within 30 days prior to the date informed consent was obtained.
14. History of alcohol or drug/abuse within 12 months prior to date informed consent was obtained.
15. Is allergic to any component of the sarilumab formulation.
16. Pregnant or breastfeeding.
17. Any condition that, in the opinion of the investigator, contraindicates participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hirsh D Komarow, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
.Human data generated in this study will be shared for future research as follows:
  * De-identified data in an NIH-funded or approved public repository.
  * De-identified data in another public repository.
  * Identified data in the Biomedical Translational Research Information System (BTRIS, automatic for activities in the CC) and the Genomic Research Integration System (GRIS).
  * De-identified or identified data with approved outside collaborators under appropriate agreements.
Time Frame: One year after submission of result
Access Criteria: Request to PI

REFERENCES:
- [Derived] Komarow HD, Wang J, Eisch R, Scott L, Brittain EH, Metcalfe DD. Treatment of indolent systemic mastocytosis with sarilumab is not supported in a randomized trial. J Allergy Clin Immunol Glob. 2025 May 21;4(3):100498. doi: 10.1016/j.jacig.2025.100498. eCollection 2025 Aug. PMID 40529483
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-I-0027.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 21 participants were enrolled in the study and five participants were deemed ineligible and excluded from study
Period: Overall Study
Arm/Group | Drug: Sarilumab | Placebo
Started | 8 | 8
Completed | 5 | 7
Not Completed | 3 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Drug: Sarilumab | Placebo | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 5 | 12
  >=65 years | 1 | 3 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 3 | 5 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 8 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 7 | 5 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Quality of Life (QoL) Using Mastocytosis Quality of Life Questionnaire (MC-QoL)
Description: The Mastocytosis Quality of Life Questionnaire (MC-QoL) is a validated health-related quality of life (QoL) survey for patients with mastocytosis that consists of 27 items and is divided into four domains: symptoms, social life/functioning, emotions, and skin. Each item has five options scored from 0-4 for a total minimum score of zero and maximum score of 108. The raw scores were transformed to a 0 to 100 scale. The overall disease impairment on QoL is measured by assessing both the total score and the scores of each domain with higher scores of 25% or greater indicating a higher QoL impairment.
  The percent change in QoL from baseline to 16 weeks post-initiation of study for participants was computed as [(Baseline QoL - 16-week QoL)/Baseline QoL] × 100]. Positive value indicates improvement.
Time Frame: Baseline and 16-week post-initiation of study
Population: Modified Intent-to-Treat (mITT) participants who completed questionnaire during the blinded phase of the study. One participant did not complete study during the blinded phase so was excluded from analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of change in quality of life
Arm/Group | Drug: Sarilumab | Placebo
Number analyzed (Participants) | 8 | 7
percentage of change in quality of life | 38.98 [28.83 to 49.13] | 33.02 [22.17 to 43.88]
Statistical Analysis 1: Comparison: Drug: Sarilumab vs Placebo; Test type: Other; p = 0.7740, Regression, Linear

2. Primary Outcome: Number of Participants With Adverse Events by Grade
Description: Severity of adverse event by grade using Terminology Criteria for Adverse Events (CTCAE) version 5.0:
  Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age appropriate instrumental activity of daily living (ADL).
  Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activity of daily living (ADL).
  Grade 4 Life-threatening consequences; urgent intervention indicated.
  Grade 5 Death related to adverse event
Time Frame: Up to 32 weeks post initiation of study
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Drug: Sarilumab | Placebo
Number analyzed (Participants) | 8 | 7
Participants
  Grade 1 | 7 | 6
  Grade 2 | 6 | 3
  Grade 3 | 2 | 2
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0

3. Secondary Outcome: Percent Change in Quality of Life (QoL) Using the Memorial Symptom Assessment Scale (MSAS)
Description: The Memorial Symptom Assessment Scale (MSAS) is used to evaluate a patient's experience with 32 symptoms over the course of the previous week. Symptoms are evaluated by severity (0 = not at all to 4 = very severe) and distress (0 = not at all to 4 = very much] for eight of the symptoms, and for severity, distress, and frequency (0 = not at all to 4 = almost constantly) for the remaining 24 symptoms for a total minimum score of zero and maximum score of 352. Higher score indicates worsening condition.
  The result is calculated by taking the average of the scores for the 32 questions for baseline and week 16 post initiation of study. The percent change in quality of life (QoL) from baseline to 16 weeks post-initiation of study for participants was computed as [(Baseline QoL - 16-week QoL)/Baseline QoL] × 100]. Positive value indicates improvement.
Time Frame: Baseline and 16-week post-initiation of study
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of change in quality of life
Arm/Group | Drug: Sarilumab | Placebo
Number analyzed (Participants) | 8 | 7
percentage of change in quality of life | 0.767 [0.54 to 0.99] | 0.503 [0.26 to 0.74]
Statistical Analysis 1: Comparison: Drug: Sarilumab vs Placebo; Test type: Other; p = 0.1071, Regression, Linear

4. Secondary Outcome: Percent Change in Quality of Life (QoL) Using Mastocytosis Quality of Life Questionnaire (MQLQ)
Description: The Mastocytosis Quality of Life Questionnaire (MQLQ) is disease specific quality of life questionnaire consisting of 49 questions to assess the effect of mastocytosis on daily life. It includes the role of mastocytosis in 8 domains: fatigue and mental health, anaphylaxis, bone symptoms, unfamiliarity (low awareness), flushing, general symptoms, skin symptoms, and triggers. Each item in the 49 questions has seven options scored from 0-6 with a minimum total score of zero and a maximum total score of 294. Higher score indicates worsening condition.
  The result is calculated by summing scores from all 49 items for baseline and week 16 post initiation of study. The percent change in QoL from baseline to 16 weeks post-initiation of study for participants was computed as [(Baseline QoL - 16-week QoL)/Baseline QoL] × 100]. Positive value indicates improvement.
Time Frame: Baseline and 16-week post-initiation of study
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of change in quality of life
Arm/Group | Drug: Sarilumab | Placebo
Number analyzed (Participants) | 8 | 7
percentage of change in quality of life | 111.02 [88.51 to 133.53] | 100.26 [76.19 to 124.33]
Statistical Analysis 1: Comparison: Drug: Sarilumab vs Placebo; Test type: Other; p = 0.4904, Regression, Linear

5. Secondary Outcome: Percent Change in Quality of Life (QoL) Using Mastocytosis Symptoms Assessment Form (MSAF)
Description: The Mastocytosis Symptoms Assessment Form (MSAF) is a 22-item questionnaire that assesses the severity of symptoms with an 11-point numeric rating scale, where "0 = No symptom" and "10 = Worst imaginable symptom" for a total minimum score of zero and total maximum score of 220. Higher score indicates worsening condition.
  The result is calculated by summing scores from all 22 items for baseline and week 16 post initiation of study. The percent change in QoL from baseline to 16 weeks post-initiation of study for participants was computed as [(Baseline QoL - 16-week QoL)/Baseline QoL] × 100]. Positive value indicates improvement.
Time Frame: Baseline and 16-week post-initiation of study
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of change in quality of life
Arm/Group | Drug: Sarilumab | Placebo
Number analyzed (Participants) | 8 | 7
percentage of change in quality of life | 55.83 [43.00 to 68.66] | 42.20 [28.48 to 55.91]
Statistical Analysis 1: Comparison: Drug: Sarilumab vs Placebo; Test type: Other; p = 0.1399, Regression, Linear

ADVERSE EVENTS:
Time Frame: Up to 16 weeks after final dose of intervention
Arm/Group | Drug: Sarilumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/8
Other Adverse Events (participants affected / at risk) | 7/8 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Drug: Sarilumab (N=8) | Placebo (N=8)
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Drug: Sarilumab (N=8) | Placebo (N=8)
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1
Dizziness (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0
Eye pain (Eye disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Pharyngitis (Gastrointestinal disorders) | 2 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Adverse reaction (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Influenza like illness (General disorders) | 1 | 0
Injection site bruising (General disorders) | 1 | 0
Injection site erythema (General disorders) | 3 | 0
Injection site induration (General disorders) | 1 | 0
Injection site reaction (General disorders) | 0 | 1
Irritability (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Procedural pain (General disorders) | 0 | 1
Bacterial vaginosis (Infections and infestations) | 1 | 0
Candida infection (Infections and infestations) | 3 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 2 | 0
Blood chloride increased (Investigations) | 0 | 1
Blood cholesterol increased (Investigations) | 2 | 0
Lymphocyte count decreased (Investigations) | 1 | 3
Neutrophil count decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 3 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Insomnia (Nervous system disorders) | 1 | 2
Memory impairment (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Sensory disturbance (Nervous system disorders) | 0 | 1
Genitourinary tract infection (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Dysmenorrhea (Reproductive system and breast disorders) | 1 | 0
Perimenopausal symptoms (Reproductive system and breast disorders) | 0 | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chest discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-18): https://cdn.clinicaltrials.gov/large-docs/73/NCT03770273/Prot_SAP_000.pdf